CLINICAL TRIAL: NCT06840028
Title: Effects of Personalized Exercise Prescriptions Through Mobile Health on Physical Activity and Health Outcomes in the Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: University of Tennessee (Other); University of Tennessee Medical Center (Other)
Responsible Party: Principal Investigator, Zan Gao, Professor and Department Head, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UTK IRB-24-07955-XP
Record Dates: First submitted 2025-02-05; First posted 2025-02-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-02

CONDITIONS: Cancer Survivors; Chronic Disease; Physical Activity; Cancer Survivorship; Physical Inactivity; Physical Activity in Adults
Keywords: U.S Cancer survivors; Tennessee Cancer Survivors; Cancer patient; Cancer; Chronic Disease; Physical Activity; Physical Inactivity; Rural oncology; Rural Health; Cancer outcomes; Cancer Recovery
MeSH Terms: conditions — Chronic Disease; Motor Activity; Sedentary Behavior; Neoplasms | interventions — Telemedicine; Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group participants would receive access to a study-developed mHealth application, sFitRx, that delivers personalized PA programming as well as be provided with a fitness tracker to monitor their habitual PA levels.
  Interventions: Other: mHealth/sFitRx
- Comparison Group (Active Comparator): Comparison Group participants would receive the fitness tracker only.
  Interventions: Other: Fitness Tracker

INTERVENTIONS:
Other: mHealth/sFitRx — Experimental Group - Will receive a personalized mHealth application and fitness tracker. Specifically, Experimental Group participants will receive the sFitRx smartphone application that provides weekly personalized PA interventions informed by big data analysis. They will also receive a Fitbit Inspire 3 to track real-time PA, with PA data uploaded to Fitabase. Importantly, the PA data from the Fitbit Inspire 3 will inform the big data analyses used to generate the personalized PA intervention provided by the sFitRx application.
  Arms: Experimental Group
Other: Fitness Tracker — Comparison Group - Will receive the Fitbit Inspire 3 only.
  Arms: Comparison Group

SUMMARY:
Participation in regular physical activity is vital to a healthy lifestyle. Research has shown that regular participation in physical activity among cancer survivors is not only able to improve health outcomes, but is also related to their quality of life.

As we live in an age of technology, health wearables and smartphone apps might be one novel manner by which to help cancer survivors increase physical activity as well as improve health outcomes. Yet, the effectiveness of wearable and app as a tool for health promotion among cancer survivors is largely unstudied.

The purpose of this study is to evaluate the effectiveness of a personalized m-health intervention via fitness wearable (Fitbit Inspire 3) exercise app (sFitRx) on physical activity, weight, quality of life, individual beliefs, and emotions among cancer survivors.

DETAILED DESCRIPTION:
Cancer remains a vital public health concern in the U.S. Research has shown that physical activity (PA) provides many physical and mental health benefits after cancer diagnosis and plays an important role in reducing all-cause and cancer-related mortality, as well as cancer incidence, in cancer survivors (CS). Adopting a physically active lifestyle is therefore crucial to decrease cancer risk and improve cancer prognosis and quality of life. However, most CS do not achieve the recommended 150 min/week of moderate-to-vigorous PA (MVPA). This issue is particularly pronounced for CS in low-income, underserved areas who tend to have considerably less access to PA-conducive environments compared to their more affluent peers. It is therefore imperative to study innovative, ease-to-implement health interventions CS that can promote increased engagement and self-regulation of health behaviors, such as PA, while also improving other health outcomes; thereby offering better supportive care.

One promising easy-to-implement medium to improve engagement in and self-regulation of health behaviors is mobile health (mHealth), which includes advanced smartphone application technology often combined with wearables and social media to improve the healthcare delivery experience. Researchers have recently applied such technologies with CS to promote improved health through increased PA and reduced sedentary behavior (SB), with observations promising. Despite promising observations, these studies were often conducted with small samples over short durations (less than or equal to three months), with the interventions lacking personalized PA prescriptions informed by back end big data analysis techniques to further improve intervention implementation. As such, examining how a longer-term tailored, big data-informed mHealth PA intervention in CS might improve health and well-being would fill a major literature gap.

The investigators thus propose a 12-month randomized-controlled trial to investigate how an mHealth-delivered PA intervention informed by big data analysis (hereafter, 'personalized mHealth intervention') can improve the health and well-being of CS over a 12-month period. Experimental Group participants would receive access to a study-developed mHealth application, sFitRx, that delivers personalized PA programming as well as be provided with a fitness tracker to monitor their habitual PA levels. Comparison Group participants would receive the fitness tracker only. Successful study completion will inform the development of effective, mHealth-delivered PA programs in CS that might guide health professionals in the initiation of such novel programs in lower-income communities with the goal of promoting PA and health in this population.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age
* Participant was previously diagnosed with stage 0-III cancer
* Participant have had one or more of the cancers of interest (e.g., breast, lung)
* Participant completed active cancer treatment at least three months prior to enrollment, with the exception of continued maintenance immunotherapy or endocrine therapy
* Participant possess basic English communication capability
* Participant do not participate in other health promotion programs
* Participant is an Android or Apple smartphone owner
* Participant is willing to participate in mHealth-delivered programs
* Participant is willing to consent and be randomized
* Participant has no contraindications to PA participation

Exclusion Criteria:

* Participant is currently undergoing chemotherapy or radiation as primary cancer treatment
* Having any contraindications that might interfere with PA engagement, such as a medical condition and pacemaker implant
* Plan to relocate or travel for >two weeks during the study period;
* Presence of distant metastasis
* Planning or preparing for surgery as primary treatment or as a reconstruction procedure in the next 3 months
* Have a stage 4 cancer diagnosis
* Participant is already engaging in ≥75 min/week of vigorous-intensity PA, ≥150 min/week of moderate-intensity PA, or an equivalent combination of both over the last 3 months
* An unstable mental condition that would prevent following study protocols
* Reporting a Physical Activity Readiness Questionnaire (PAR-Q) score that indicates PA may be unsafe
* Being a prisoner, pregnant, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Baseline (i.e., pre-intervention), six months, and 12 months.
  Physical Activity. CS's mean steps/day will be the primary outcome and will be assessed using Fitbit Inspire. Participants will be instructed to wear the Fitbit on the non-dominant wrist at all times throughout the study.

SECONDARY OUTCOMES:
Health Indicators | Baseline (i.e., pre-intervention), six months, and 12 months.
  Participants' height (m) and weight (kg) will be measured at home by themselves, with body mass index (BMI) calculated by their height and weight (kg/m^2).43
Health Indicators | Baseline (i.e., pre-intervention), six months, and 12 months.
  Psychosocial beliefs (e.g., self-efficacy, social support) will be assessed by standardized self-report surveys through established questionnaires.45-50
Health Indicators | Baseline (i.e., pre-intervention), six months, and 12 months.
  The investigators will assess quality of life (QoL) using the Patient Reported Outcome Measurement Information System44. Investigators are most interested in assessing physical functioning, anxiety, and depression.
Physical Activity | Baseline (i.e., pre-intervention), six months, and 12 months.
  Mean calories burned/day and SB/day will also be examined as a secondary outcome. As mentioned previously, investigators will retrieve Fitbit data via Fitabase.40-42
Health Indicators | Baseline (i.e., pre-intervention), six months, and 12 months.
  The researchers will assess participants emotions via the Positive and Negative Affect Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided